CLINICAL TRIAL: NCT01057147
Title: A Phase II, Prospective, Randomized, Double-masked, Parallel Group, Multi-center Study Assessing the Safety and Efficacy of 2% Rebamipide (OPC-12759) Compared to Placebo in Clearing of Fluorescein Staining of the Central Cornea in Subjects With Keratoconjunctivitis Sicca (Dry Eye)
Brief Title: Safety and Efficacy Study of Rebamipide 2% Ophthalmic Suspension in Subjects With Dry Eye - Effects on Central Cornea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU-RED-204
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Keratoconjunctivitis Sicca; Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- rebamipide 2% ophthalmic suspension (Experimental)
  Interventions: Drug: rebamipide 2% ophthalmic suspension
- placebo eye drops (Placebo Comparator)
  Interventions: Drug: placebo eye drops

INTERVENTIONS:
Drug: rebamipide 2% ophthalmic suspension — Instill one drop in each eye four times daily for 12 weeks.
  Arms: rebamipide 2% ophthalmic suspension
Drug: placebo eye drops — Instill one drop in each eye four times daily for 12 weeks.
  Arms: placebo eye drops

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 2% rebamipide compared to placebo in clearing of fluorescein staining of the central cornea in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of dry eye as defined by the protocol
* Central corneal staining

Exclusion Criteria:

* Ongoing ocular disease that may interfere with study parameters
* Inability to stop using topical ophthalmic medications throughout the duration of the study
* Inability to stop the use of contact lenses for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Central corneal clearing as measured by fluorescein staining | 12 weeks

SECONDARY OUTCOMES:
Ocular staining | 12 weeks
Dry eye symptoms | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Kubota, MD, PhD, Study Director — Kubota Vision Inc.
Locations (19):
- United States (19):
  - East Valley Ophthalmology, Mesa, Arizona
  - Arizona Center for Clinical Trials, LLC, Phoenix, Arizona
  - Cornea Consultants of Arizona, Phoenix, Arizona
  - Macy Eye Center, Los Angeles, California
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Specialty Eye Care, Parker, Colorado
  - Cohen Laser and Vision Center, Boca Raton, Florida
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Med Eye Associates, Miami, Florida
  - George R. John, MD, Louisville, Kentucky
  - Central Maine Eye Care, Lewiston, Maine
  - Ora, Inc., Andover, Massachusetts
  - Ophthalmology Associates, St Louis, Missouri
  - Nevada Eye Care Professionals, Las Vegas, Nevada
  - Avista Eye Center, Las Vegas, Nevada
  - New York Ophthalmology, PC, Manhasset, New York
  - Mundorf Eye Center, Charlotte, North Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - The Cataract & Glaucoma Center, El Paso, Texas